CLINICAL TRIAL: NCT01599338
Title: Influence du Victoza (Liraglutide,Analogue GLP-1) Sur Les Performances Gustatives, le Rassasiement Sensoriel spécifique, le Liking et le Wanting Chez Les Patients diabétiques de Type 2.
Brief Title: Impact of Liraglutide on Sensory Perception, Sensory Specific Satiety, Liking and Wanting in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Marie Claude Brindisi, MD, Centre Hospitalier Universitaire Dijon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: A100991-10; 2010-022618-19 (EudraCT Number)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus; Overweight
Keywords: Liraglutide; GLP-1 analogue; Food preference; Gustative perception; Liking; wanting; T2DM; body mass composition; leptin; ghrelin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Food Preferences | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liraglutide (Experimental): Single Arm study. T2DM patients are studied before and after 3 months of Liraglutide treatment (1.2 mg/day).
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — 3 months of treatment by Liraglutide (self-administration). The initial dose was 0.6 mg/day subcutaneously during five days, then uptitrated to a daily dose of 1.2 mg during three months.
  Other Names: Novonordisk (Puteaux, France)

SUMMARY:
Besides their potential action in the treatment of type 2 diabetes mellitus (T2DM), GLP-1 analogues decrease satiety and food intake leading to a significant weight loss in patients. However, little is known about their effects on food hedonic sensations and taste perception.

The aim of this study is to investigate the impact of Liraglutide on the liking and wanting components of the food reward system, taste sensitivity and sensory specific satiety in type 2 diabetes mellitus (T2DM) patients. According to the review of literature in animal models, it is expected that Liraglutide will modify food preference and gustative perception in humans.

Thirty T2DM patients will be studied before and after 3 months of treatment with Liraglutide (1.2 mg/day). Same tests will be carried out on two consecutive days before and after the treatment administration. Olfactory liking, recalled liking and wanting for several food items will be assessed. Sensory specific satiety will be measured as well as detection thresholds for salty, sweet and bitter tastes. Subjects will also answer questionnaires on hunger, pleasure in eating, and food intake.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetic patients

1. with glycemic unbalance despite anti-diabetic treatments and
2. overweight (BMI > 25 kg/m²)

Exclusion Criteria:

* Impaired renal function (creatinine clearance < 50 ml/min),
* Pregnancy,
* Congestive heart failure,
* Acute and chronic infection,
* Evolutive cancer,
* Cirrhosis,
* Ongoing antibiotic treatment,
* Smoking (more than 5 cig/day),
* Alcohol consumption (more than 20 g/day),
* Aversion for the foods eaten or smelt during the study,
* Impaired comprehension for cognitive tasks,
* Treatments known to interfere with olfactory and gustative performances

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in liking and wanting for protein, lipid and glucid foods | 3 months
Change in sensory specific satiety for protein, lipid and glucid foods | 3 months
Change in gustative detection thresholds for sweet, bitter and salty tastes | 3 months
Change in appetite, desire to eat, pleasure in eating | 3 months

SECONDARY OUTCOMES:
Change in body mass composition (Dual Energy XRay Absorptiometry) | 3 months
Change in plasma ghrelin, leptin, and HbA1c levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Brindisi, MD, Principal Investigator — CHU Dijon
Locations (1):
- CHU Dijon, Dijon, Bourgogne-Franche-Comté, France